CLINICAL TRIAL: NCT00386139
Title: An Eight-week Multicenter Study to Evaluate the Efficacy and Safety of the Combination of Aliskiren / HCTZ (300/12.5 mg and 300/25 mg) in Comparison With Aliskiren 300 mg in Patients With Essential Hypertension Not Adequately Responsive to Aliskiren 300 mg Monotherapy
Brief Title: A Safety and Efficacy Trial of the Combination of Aliskiren / Hydrochlorothiazide (HCTZ)(300/12.5 mg and 300/25 mg) Compared to Aliskiren 300 mg in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2332
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: Diastolic; systolic; hypertension; aliskiren; blood pressure; hydrochlorothiazide, HCTZ
MeSH Terms: conditions — Hypertension; Heart Murmurs; Systolic Murmurs

INTERVENTIONS:
Drug: Aliskiren/HCTZ

SUMMARY:
Evaluate the diastolic blood pressure lowering effect of combination of aliskiren 300 mg and HCTZ (12.5 mg and 25 mg) in hypertensive patients who do not show sufficient blood pressure response to aliskiren 300 mg.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18 years old or older.
* Patients with a diagnosis of hypertension.
* Patients who are eligible and consent to participate in the study

Exclusion Criteria:

* Severe hypertension
* Previous or current diagnosis of heart failure.
* History of hypertensive encephalopathy or cerebrovascular accident, transient ischemic cerebral attack (TIA), myocardial infarction, coronary bypass surgery, or any percutaneous coronary intervention (PCI).
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 881 (Actual)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Mean Sitting Diastolic Blood Pressure lowering effect at baseline, and week 8.

SECONDARY OUTCOMES:
Mean sitting systolic blood pressure (msDBP) lowering from baseline to week 8
Safety and tolerability
Proportion of patients achieving a blood pressure control target at week 8

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Result] Nickenig G, Simanenkov V, Lembo G, Rodriguez P, Salko T, Ritter S, Zhang J. Efficacy of aliskiren/hydrochlorothiazide single-pill combinations in aliskiren non-responders. Blood Press Suppl. 2008 Dec;2:31-40. doi: 10.1080/08038020802507290. PMID 19203020